CLINICAL TRIAL: NCT05927116
Title: A Mobile Phone App-based Intervention for Supporting and Empowering Parents of Children With Autism Spectrum Disorder (ASD): a Randomised Waitlist-controlled Trial
Brief Title: RCT of a Mobile Phone App-based Intervention for Parents of Children With Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Wing Ho, Assistant Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022.584; 10210356 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2023-06-04; First posted 2023-07-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Parent-Child Relations
Keywords: digital interventions; parenting; mindfulness; psychoeducation
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomised wait-list controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): Both groups will be assessed at baseline on the outcome measurements, after which the immediate intervention group will begin the 6-week intervention
  Interventions: Other: Mobile phone app-based intervention for supporting and empowering parents of children with autism spectrum disorder (ASD)
- Waitlist control (No Intervention): Both groups will be assessed at baseline on the outcome measurements, after which the the waitlist control group will receive usual care in the following six weeks. Afterwards, the waitlist control group will complete outcome assessment once again, before receiving the 6-week intervention

INTERVENTIONS:
Other: Mobile phone app-based intervention for supporting and empowering parents of children with autism spectrum disorder (ASD) — TRIP is a mobile app-based intervention comprises of a 6-week structured training on mindfulness and educational modules on ASD parenting skills.
  Other Names: TRIP app for ASD parents
  Arms: Immediate intervention

SUMMARY:
The objective of this study is to evaluate the effectiveness of a 6-week mobile app-based intervention in empowering and supporting Chinese parents of ASD children through knowledge and skills transfer and mindfulness training, to explore factors associated with enhanced user experiences and sustained usage through participants' qualitative feedback and observing naturalistic usage patterns beyond the active intervention period, and to refine the mobile app based on the data prior to wider dissemination of the app. We hypothesise that there will be a greater reduction in parental stress and mood symptoms, and improvement of mindfulness attitude and parenting competence in parents with ASD children after the 6-week app-based intervention than the waitlist controls.

DETAILED DESCRIPTION:
Parents of autism spectrum disorder (ASD) children are often stressed about challenges in raising their children with multifaceted needs, and their stress could undermine the child's development. With the ever-increasing demand in clinical services and disruptions by coronavirus pandemic (COVID-19), we aim to investigate the clinical efficacy of a mobile app-based intervention in reducing stress and mood symptoms, and enhancing mindfulness and competence in parents of children with ASD. The 6-week mobile app-based intervention programme is a structured course of mindfulness training, and knowledge and skills transfer of parenting ASD children with specific content personalised to the participant's needs, which was developed as an accessible and scalable primary-level care platform to improve the well-being of parents.

In this study, a pragmatic, randomized waitlist-controlled trial will be conducted. 700 parents of ASD children who are ≤12 years of age and either 1. waiting for, or 2. actively receiving treatment from a regional children psychiatric specialist clinic will be recruited. Parents will be randomized into an immediate intervention arm and a waitlist arm. Parental stress level, mood symptoms, competence, and level of mindfulness will be measured before, immediately after, and 2 months after the intervention with self-reported questionnaires. Outcome measurement of pre- and post-intervention from the two groups of participants will be analysed with a Mixed Factorial ANOVA. A treatment x time effect on the outcome measurement is expected.

The results of the proposed study will provide evidence to the real-life efficacy of a mobile app-based intervention service model to support parents of children with ASD in the era of digital mental health. As the impact of mental well-being of parents extends beyond the parents themselves, effective management of the elevated level of parental stress in ASD families is beneficial to the family functioning and long-term development of the child. The solid evidence from this sizable clinical trial can also inform clinicians and service-users in choosing the evidence-based intervention suitable to their context, among the range of commercially available products with claimed efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Chinese parents living in Hong Kong
* Parents caring for ASD children, diagnosed by clinicians according to the criteria of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria and aged ≤12
* Recruited from the Child and Adolescent Psychiatric clinic at the Alice Ho Miu Ling Nethersole Hospital, a regional hospital providing the sole public child and adolescent psychiatric service in the New-Territory East Cluster of the Hospital Authority in Hong Kong
* Able to read and understand Cantonese
* Have access to an internet-enabled mobile phone with a valid phone number for the duration of the trial

Exclusion Criteria:

* Parents who are not the main carer of their ASD children
* Currently receiving psychological interventions
* Undergoing mindfulness training will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Parental anxiety | Pre-intervention
  Measured by the 7-item Generalised Anxiety Disorder scale (GAD-7; Spitzer et al., 2006) for anxiety symptoms. GAD-7 scores range from 0 to 21, higher scores indicating greater levels of anxiety symptoms.
Parental anxiety | Immediately post-intervention
  Measured by the 7-item Generalised Anxiety Disorder scale (GAD-7; Spitzer et al., 2006) for anxiety symptoms. GAD-7 scores range from 0 to 21, higher scores indicating greater levels of anxiety symptoms.
Parental anxiety | 2-months post-intervention
  Measured by the 7-item Generalised Anxiety Disorder scale (GAD-7; Spitzer et al., 2006) for anxiety symptoms. GAD-7 scores range from 0 to 21, higher scores indicating greater levels of anxiety symptoms.
Parental depression | Pre-intervention
  Measured by the 9-item Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) for depressive symptoms. PHQ-9 scores range from 0 to 27, higher scores indicating greater levels of depressive symptoms.
Parental depression | Immediately post-intervention
  Measured by the 9-item Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) for depressive symptoms. PHQ-9 scores range from 0 to 27, higher scores indicating greater levels of depressive symptoms.
Parental depression | 2-months post-intervention
  Measured by the 9-item Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) for depressive symptoms. PHQ-9 scores range from 0 to 27, higher scores indicating greater levels of depressive symptoms.
Parenting stress | Pre-intervention
  Measured by the 36-item Parenting Stress Index-Short Form (PSI-SF), considering three domains of parenting distress, difficult child, and parent-child dysfunctional interaction. Scores range from 36 to 180, with higher scores indicating greater levels of stress.
Parenting stress | Immediately post-intervention
  Measured by the 36-item Parenting Stress Index-Short Form (PSI-SF), considering three domains of parenting distress, difficult child, and parent-child dysfunctional interaction. Scores range from 36 to 180, with higher scores indicating greater levels of stress.
Parenting stress | 2-months post-intervention
  Measured by the 36-item Parenting Stress Index-Short Form (PSI-SF), considering three domains of parenting distress, difficult child, and parent-child dysfunctional interaction. Scores range from 36 to 180, with higher scores indicating greater levels of stress.
Parenting competence | Pre-intervention
  Measured by the 17-item Parenting Sense of Competence scale (PSOC; Gibaud-Wallston & Wandersman, 1978). Scores ranges between 17 to 102, with higher scores indicating a higher parenting sense of competency.
Parenting competence | Immediately post-intervention
  Measured by the 17-item Parenting Sense of Competence scale (PSOC; Gibaud-Wallston & Wandersman, 1978). Scores ranges between 17 to 102, with higher scores indicating a higher parenting sense of competency.
Parenting competence | 2-months post-intervention
  Measured by the 17-item Parenting Sense of Competence scale (PSOC; Gibaud-Wallston & Wandersman, 1978). Scores ranges between 17 to 102, with higher scores indicating a higher parenting sense of competency.
Parenting efficacy | Pre-intervention
  Measured by the 6-item Parenting Efficacy subscale of the Parenting Self-Agency Measure (Dumka et al., 1996). Scores ranges between 6-42, with higher scores indicating higher levels of parenting efficacy.
Parenting efficacy | Immediately post-intervention
  Measured by the 6-item Parenting Efficacy subscale of the Parenting Self-Agency Measure (Dumka et al., 1996). Scores ranges between 6-42, with higher scores indicating higher levels of parenting efficacy.
Parenting efficacy | 2-months post-intervention
  Measured by the 6-item Parenting Efficacy subscale of the Parenting Self-Agency Measure (Dumka et al., 1996). Scores ranges between 6-42, with higher scores indicating higher levels of parenting efficacy.

SECONDARY OUTCOMES:
App usability | Immediately post-intervention
  Measured by the 10-item System Usability Scale (SUS; Brooke, 1996) for assessing the usability of products and apps. SUS scores have a range of 0 to 100, with a higher score means greater app usability.
App satisfaction | Immediately post-intervention
  App satisfaction will be measured by open-ended questions regarding suggestions for improvement of the app, for the purpose of refinement of the app.
Number of app usage days beyond the 6-week structured intervention | 6-months post-intervention
  Number of days with logins beyond the 6-week intervention period
Average duration of app usage beyond the 6-week structured intervention | 6-months post-intervention
  Time spent in app per login beyond the 6-week intervention period
Number of mindfulness practices completed beyond the 6-week structured intervention | 6-months post-intervention
  Number of guided mindfulness sessions beyond the 6-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Wong, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No